CLINICAL TRIAL: NCT03984994
Title: Increasing Muscle Capillarization to Enhance Responses to Strength Training in Sarcopenia
Brief Title: Muscle Capillarization and Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: University of Maryland, Baltimore (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Steven J. Prior, Ph.D., Assistant Professor, University of Maryland, College Park
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00086001; 5R21AG064571 (NIH)
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Sarcopenia
Keywords: muscle; capillary; exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The study employs 2 interventions: resistance training and aerobic exercise training. One group of participants will undergo resistance training then aerobic exercise training; the other group will undergo aerobic exercise training then resistance training.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise training followed by resistance training (Experimental): Participants in this arm will undergo 3 months of aerobic exercise training, followed by 3 months of strength training
  Interventions: Other: Aerobic exercise training; Other: Strength training
- Resistance training followed by aerobic exercise training (Active Comparator): Participants in this arm will undergo 3 months of strength training, followed by 3 months of aerobic exercise training
  Interventions: Other: Aerobic exercise training; Other: Strength training

INTERVENTIONS:
Other: Aerobic exercise training — 3 months of center-based, supervised treadmill exercise
Other: Strength training — 3 months of center-based, supervise strength training

SUMMARY:
Aging is associated with a loss of muscle mass, termed sarcopenia, that reduces mobility, decreases physical function and accelerates progression of other age-related disorders. This study is designed to determine whether increasing skeletal muscle capillarization through aerobic exercise will enhance muscular adaptations to strength training in older adults with sarcopenia.

DETAILED DESCRIPTION:
Sarcopenia, or the aging-related loss of muscle mass, affects a large number of older adults. The presence of sarcopenia is associated with physical disability, poor quality of life, and all-cause mortality, in part because sarcopenic adults have low muscle skeletal muscle capillarization and may lack the adequate perfusion needed to maintain muscle mass and function. This study will test the effects of increasing skeletal muscle capillarization through aerobic exercise training on responses to resistance training in older adults. Eligible participants will be randomized to one of two groups, resistance training preceded by aerobic exercise training (AEX-RT), or resistance training followed by aerobic exercise training (RT-AEX). Participants in the AEX-RT group will undergo 3 months of aerobic exercise training to increase skeletal muscle capillarization, followed by 3 months of resistance training. Participants in the RT-AEX group will undergo 3 months of resistance training, followed by 3 months of aerobic exercise training. Before and after the interventions, participants will undergo assessments of muscle size, strength, and capillarization, as well as assessments of physical function.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index = 18-32.5 kg/m2
* Non-smoker
* Presence of at least moderate sarcopenia (low muscle mass per unit body height)

Exclusion Criteria:

* Diagnosis of diabetes, cancer, pulmonary or renal disease
* Physical impairment preventing exercise
* Recent history of exercise training

Ages: 65 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, Baltimore & Baltimore VA Medical Center, Baltimore, Maryland
  - University of Maryland, College Park, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants are assigned to groups upon completion of baseline testing.
Period: Overall Study
Arm/Group | Aerobic Exercise Training Followed by Resistance Training | Resistance Training Followed by Aerobic Exercise Training
Started | 7 | 7
Completed | 5 | 6
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: All participants assigned to an intervention are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise Training Followed by Resistance Training | Resistance Training Followed by Aerobic Exercise Training | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (4) | 73 (6) | 75 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
Appendicular Lean Mass (kg) [Mean (Standard Deviation); unit: kilograms] | 17.1 (1.9) | 19.3 (5.4) | 18.4 (4.4)
Quadriceps muscle strength (Newton*meters) [Mean (Standard Deviation); unit: Newton*meters] | 91 (15) | 107 (30) | 101 (25)

OUTCOME MEASURES:

1. Primary Outcome: Skeletal Muscle Capillarization
Description: Change in the number of capillaries per unit of skeletal muscle tissue after resistance training. The aims of the study were to compare responses to resistance training between arms/groups. Therefore, only the resistance training-induced change (post minus pre-resistance training) is assessed and analyzed as this is the primary outcome for each arm.
Time Frame: 3 months (post minus pre-resistance training)
Population: All participants completing the resistance training portion of the intervention in each arm were analyzed. Only data for the resistance training portion of the study are reported (change post-pre training). Data and analyses are not reported for aerobic exercise as this was not part of the aims/outcomes and was only assessed to gauge responses to only RT.
Measure: Mean (Standard Error); unit: capillaries per muscle fiber
Arm/Group | Aerobic Exercise Training Followed by Resistance Training | Resistance Training Followed by Aerobic Exercise Training
Number analyzed (Participants) | 5 | 6
capillaries per muscle fiber | 0.4 (0.1) | 0.2 (0.1)
Statistical Analysis 1: Comparison: Aerobic Exercise Training Followed by Resistance Training vs Resistance Training Followed by Aerobic Exercise Training; Per the aims of the study, the responses to RT were compared between 2 arms/groups. The change in the outcome (post-RT minus pre-RT) in each arm/group was compared using a t-test. Responses to AEX training itself are not assessed as this was not an aim or hypothesis of the study. The hypothesis was that the "Aerobic exercise training followed by resistance training" arm would have greater changes/improvements in study outcomes than the "Resistance training followed by aerobic training" group; Test type: Superiority; p = 0.27, t-test, 2 sided; Mean Difference (Final Values) = 0.2

2. Primary Outcome: Quadriceps Muscle Cross-sectional Area
Description: Change in the size of the thigh muscles. The aims of the study were to compare responses to resistance training between arms/groups. Therefore, only the resistance training-induced change (post minus pre-resistance training) is assessed and analyzed as this is the primary outcome for each arm.
Time Frame: 3 months (post minus pre-resistance training)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: square centimeters
Arm/Group | Aerobic Exercise Training Followed by Resistance Training | Resistance Training Followed by Aerobic Exercise Training
Number analyzed (Participants) | 5 | 6
square centimeters | 2.5 (2.0) | 0.7 (2.6)
Statistical Analysis 1: Comparison: Aerobic Exercise Training Followed by Resistance Training vs Resistance Training Followed by Aerobic Exercise Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.22, t-test, 2 sided; Mean Difference (Final Values) = 1.8

3. Secondary Outcome: Skeletal Muscle Fiber Size
Description: Change in the cross-sectional size of individual thigh skeletal muscle fibers. The aims of the study were to compare responses to resistance training between arms/groups. Therefore, only the resistance training-induced change (post minus pre-resistance training) is assessed and analyzed as this is the primary outcome for each arm.
Time Frame: 3 months (post minus pre-resistance training)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: square micrometers
Arm/Group | Aerobic Exercise Training Followed by Resistance Training | Resistance Training Followed by Aerobic Exercise Training
Number analyzed (Participants) | 5 | 6
square micrometers | 607 (108) | 356 (227)
Statistical Analysis 1: Comparison: Aerobic Exercise Training Followed by Resistance Training vs Resistance Training Followed by Aerobic Exercise Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = 251

4. Secondary Outcome: Muscle Strength
Description: Change in the strength/force produced by skeletal muscles of the thigh. Only the resistance training-induced change (post minus pre-resistance training) is reported as this is the primary outcome for each arm.
Time Frame: 3 months (post minus pre-resistance training)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Newton-meters
Arm/Group | Aerobic Exercise Training Followed by Resistance Training | Resistance Training Followed by Aerobic Exercise Training
Number analyzed (Participants) | 5 | 6
Newton-meters | 12.7 (2.3) | 2.0 (5.8)
Statistical Analysis 1: Comparison: Aerobic Exercise Training Followed by Resistance Training vs Resistance Training Followed by Aerobic Exercise Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.28, t-test, 2 sided; Mean Difference (Final Values) = 10.7

ADVERSE EVENTS:
Time Frame: Data were collected over 6 months of study participation
Description: The study adhered to clinicaltrials.gov definitions.
Arm/Group | Aerobic Exercise Training Followed by Resistance Training | Resistance Training Followed by Aerobic Exercise Training
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT03984994/Prot_SAP_000.pdf